CLINICAL TRIAL: NCT01780051
Title: An Open-label, Randomized, Single-dose, 2-way Crossover Trial to Compare the Pharmacokinetics of Repaglinide2mg and MetforminHCl 500mg Complex to Combination Preparation of Repaglinide 2mg and MetforminHCl 500mg in Healthy Male Volunteers.
Brief Title: A Pharmacokinetic Study to Compare Co-administration of Repaglinide and Metformin HCl to Administration of Combination Preparation of Those Two Components
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dalim BioTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RM0818-01
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — repaglinide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: Repaglinide/Metformin combination, Repaglinide, Metformin
- Sequence B (Experimental)
  Interventions: Drug: Repaglinide/Metformin combination, Repaglinide, Metformin

INTERVENTIONS:
Drug: Repaglinide/Metformin combination, Repaglinide, Metformin — Co-administration of Repaglinide 2mg and Metformin HCl 500mg at once in period 1.
  Administration of the Combination tablet of Repaglinide 2mg/Metformin HCl 500mg) in period 2.
  Arms: Sequence A
Drug: Repaglinide/Metformin combination, Repaglinide, Metformin — Administration of the Combination tablet of Repaglinide 2mg/Metformin HCl 500mg) in period 1.
  Co-administration of Repaglinide 2mg and Metformin HCl 500mg at once in period 2.
  Arms: Sequence B

SUMMARY:
This is a phase-1, single center, open-label, randomized, single-dose, 2-way crossover study. The objective of the study is to compare the pharmacokinetic properties after co-administration of Repaglinide 2mg and Metformin hydrochloride 500mg with administration of combination preparation of Repaglinide 2mg and Metformin hydrochloride 500mg in 50 healthy male volunteers.

DETAILED DESCRIPTION:
This is a phase-1, single center, open-label, randomized, single-dose, 2-way crossover study. The objective of the study is to compare the pharmacokinetic properties after co-administration of Repaglinide 2mg and Metformin hydrochloride 500mg with administration of combination preparation of Repaglinide 2mg and Metformin hydrochloride 500mg in 50 healthy male volunteers.

* All the subjects should be admitted one day prior to scheduled study date until 4pm to Chonbuk National University Hospital Clinical Trial Center and they will be served with the same dinner. After dinner, they should keep fast, they are just allowed to drink water until 8am of the study date.

  * According to the randomly designated order, all subjects will be administrated with the study or reference products with 240mL of water at 9am(±2hours) on the first date of the study. The study or the reference products should be swallowed completely, and not to be chewed before swallowing.

    * Study product : Repanorm M 2/500mg (Dalim BioTech Co., Ltd.)
    * Reference products : Metformin HCl 500mg tablet, Repaglinide 2mg tablet

      * Subjects have to fast for 4 hours post administration of the study or reference drugs(water intake is not allowed for 1 hour before and after the administration), and should follow standardized lunch after four hours and dinner 9 hours later from the time of administration

        * Assessment and laboratory test will be performed in accordance with schedule written on the protocol

          * After having 7 days of withdrawal period, the 2nd study period will be done at 9am(±2hours). In contrast of the 1st period, Sequence B which received the study product in 1st period will take the reference drugs for the 2nd period, while the group Sequence A which received reference drugs will take the study drug. The steps of administration of drugs and process of tests are the same with the 1st period

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers ages between 20 and 55 years at screening
2. Subject with Body Mass Index(BMI) with the range of 17.5 to 30.5kg/m2 and body weight over 45kg
3. Signed informed consent with the date of signature
4. With ability to comply with all the scheduled visits, treatment plans; laboratory tests and other processes.

Exclusion Criteria:

1. Positive of blood, kidney, endocrine, lung, gastro-intestinal, cardiovascular, hepatic, psychiatric, nervous, allergy; or with past and present disease history or symptoms that are clinically significant.
2. Any conditions that are likely to affect drug absorption. ex) gastrectomy
3. Positive on urine drug tests
4. History of drinking alcohol more than 12 ounces(360mL) of beer, 1.5 ounces(45mL) of liquor; or 21 drinks/week(1drink = 5 ounces(150mL) of wine ) 6months prior to screening
5. Participation in any other clinical studies within 2months prior to scheduled study drug administration
6. With Blood pressure of ≥ 160 mmHg(Systolic blood pressure) or ≥ 90 mmHg(Diastolic blood pressure) in sitting position at screening time.
7. History of any serious substance or alcohol abuse within one year prior to screening
8. Use of any drugs known to significantly induce or inhibit drug metabolizing enzyme within 30days prior to scheduled study drug administration
9. Cigarette smoking of over 20 sticks per day.
10. Use of any prescription drugs or any over the counter drugs within 10days or quintuple half life(whichever is longer) prior to scheduled study drug administration
11. Donation of whole blood within 2months or any blood products within 1month, prior to scheduled study drug administration
12. Disability to comply with the guidelines written on the protocol
13. Severe acute/chronic medical, physical disorder or laboratory test abnormality that are likely to alter the study result and increase the risk by participating in the study and study drug administration
14. Hypersensitivity to chief component or excipient of Repaglinide
15. History of hypersensitivity to Metformin or Biguanide class of drugs
16. With renal failure or renal inadequacy caused by cardiovascular shock, acute myocardial infarction and sepsis
17. With Congestive heart failure and undergoing drug treatment.
18. Patients undergoing radioactive iodine uptake tests, such as intravenous urography, intravenous cholangiography, angiography, computed tomography using radioactive iodine
19. Patients with type 1 diabetes, acute or chronic metabolic acidosis including diabetic ketoacidosis associated with or without coma
20. With serious infection or trauma
21. Malnutrition, starvation; weakness; pituitary insufficiency or adrenal insufficiency
22. Patients with hepatic failure, pulmonary infarction, serious pulmonary dysfunction, or other conditions associated with hypoxemia, alcohol abuser, or dehydration, diarrhea; vomiting and gastro-intestinal disease
23. Proven to be unsuitable to participate in this clinical study by an investigator

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
AUCt and Cmax of repaglinide and metformin | Before study drug administration(0h) and after 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h of study drug administration.

SECONDARY OUTCOMES:
AUC∞, Tmax, t1/2, CL/F and Vd/F of repaglinide and metformin | Before study drug administration(0h) and after 0.25h, 0.5h, 0.75h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h of study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, doctor, Principal Investigator — Chounbuk National University Hospital
Locations (1):
- Chounbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea